CLINICAL TRIAL: NCT01375335
Title: The Effects of Dobutamine on Postoperative Systolic Deformation and Diastolic Function in Patients With Hypertrophic Cardiomyopathy Operated for Aortic Valve Stenosis
Brief Title: The Effects of Dobutamine on Postoperative Cardiac Function in Aortic Valve Replacement
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient patient eligible for recruitment
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1818
Record Dates: First submitted 2011-06-14; First posted 2011-06-17 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Heart Failure
Keywords: Postoperative; Dobutamine; Inotropes; Stunning; Heart failure
MeSH Terms: conditions — Heart Failure | interventions — Dobutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dobutamine (Experimental)
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Dobutamine — 90 minutes of infusion 5 ug/kg/minute followed by isotonic saline for the same duration. The sequence of the above is randomized

SUMMARY:
The use of dobutamine in postoperative hemodynamic treatment is widespread despite seemingly intact contraction of the heart. This study aims to elucidate the efficacy of low-dose dobutamine infusion in patients in the postoperative phase replacement of the aortic valve.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years
* Left ventricular posterior wall =/>12mm
* Ejection fraction > 45%
* Sinus rhythm
* Eligible for aortic valve replacement

Exclusion Criteria:

* Need for concomitant cardiac bypass operation.
* Moderate or severe insufficiency of the mitral valve
* Active endocarditis
* Insufficient ultrasound window
* Using B-blockers
* Liver insufficiency
* Patients treated with COMT-inhibitors
* Allergy towards dobutamine
* Pregnancy
* Women of fertile age who do not use relevant anti-conception
* Lacking participant consent

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cardiac output | From 0 to 90 minutes after drug initiation
  Change in cardiac output (l/min) from initiation of study drug or placebo until 90 minutes of infusion.

SECONDARY OUTCOMES:
Mean pulmonary artery pressure | From 0 to 90 minutes after drug initiation.
  Changes in pulmonary artery pressure (mmHg) from start of study drug or placebo infusion until 90 minutes after the start.
Echocardiography | From 0 minutes to 90 minutes after drug initiation
  Echocardiographic measures of systolic and diastolic heart function.
Changes in mixed venous saturation | From 0 minutes to 90 minutes after drug initiation
  Changes in mixed venous saturation (in per cent) from baseline until the end of dobutrex or placebo infusion.
norepinephrine requirement | From 0 minutes to 90 minutes after drug initiation
  The amount of norepinephrinem(mg) required to maintain adequate systemic blood pressure during the infusion period of dobutrex and placebo
Central venous pressure | From 0 minutes to 90 minutes after drug initiation
  Changes in CVP from baseline until 90 minutes of study drug or placebo infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Sloth, Professor, Study Chair — Department of Anaesthesia & Intensive Care, Århus Univerisity Hospital
Locations (1):
- Department of Anaesthesia & Intensive Care, Århus University Hospital, Aarhus, Denmark